CLINICAL TRIAL: NCT06436612
Title: Phase II Study of Magnetic Resonance Image and Computed Tomography-Guided Stereotactic Body Radiation Therapy for Abdominopelvic Sarcomas (MARS Trial)
Brief Title: Study of Magnetic Resonance Image and Computed Tomography-Guided Stereotactic Body Radiation Therapy for Abdominopelvic Sarcomas (MARS Trial)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 23-001583; NCI-2024-04364 (Registry Identifier: Clinical Trials Reporting Program)
Record Dates: First submitted 2024-05-14; First posted 2024-05-31 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-06

CONDITIONS: Abdominopelvic Sarcomas

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Arm I (Experimental): MRI or CT-guided SBRT will be delivered in the pre-operative setting. Patients will receive 5.0-6.0 Gy x 5 fractions delivered daily.
  Interventions: Radiation: Magnetic Resonance Image and Computed Tomography-Guided Stereotactic Body Radiation Therapy

INTERVENTIONS:
Radiation: Magnetic Resonance Image and Computed Tomography-Guided Stereotactic Body Radiation Therapy — stereotactic body radiation therapy (SBRT) administered over 5 days x 5.0 - 6.0 Gy for patients with abdominopelvic sarcomas.
  Other Names: Pre-operative stereotactic body radiation therapy (SBRT)

SUMMARY:
Recent advances in radiation treatment have allowed for higher doses per treatment to be delivered safely. This study plans to use an MRI-guided linear accelerator to deliver the radiation treatment to ensure that the radiation dose is administered to the cancerous tumor, not the vital body organs.

Potential participants with a sarcoma diagnosis will be referred to Radiation Oncology during this study. If the participant is interested in participating in this study, s/he receives radiation treatment daily for 5 consecutive days except for weekends and holidays. Within 12 weeks of completing the radiation therapy, the participant will have the primary tumor surgically removed. The radiation oncology team will follow the patients for 5 years after completing radiation therapy.

DETAILED DESCRIPTION:
Each patient will undergo radiation simulation and planning. A custom vac-lok bag, alpha cradle, or equivalent immobilization device will be used. Both CT and MRI simulation will be obtained, which is standard of care for any patient undergoing radiation therapy for soft tissue sarcomas.

The study investigator will be responsible for delineating the gross tumor volume (GTV) using the CT as well as MRI performed as part of staging. Guidelines for contouring will be as per the currently open NRG trial for sarcomas. In general, this may entail expansions by 5-15 mm isotropically, should include any suspicious areas be identified on T2 weighted MRI, and should be cropped to natural anatomic borders. This clinical target volume (CTV) will then be expanded to a planning treatment volume (PTV) using a 3-5 mm expansion.

A prescription dose of 5-6 Gy x 5 fractions (25-30 Gy) will be delivered to at least 95% of the PTV. Stereotactic body radiotherapy (SBRT) and/or intensity modulated radiotherapy (IMRT) planning techniques may be used to minimize radiation dose to nearby organs at risk (OAR) but is not required.

Delineation of normal structures will be performed and verified by the responsible study investigator. The radiation physicist or dosimetrist will optimize the treatment plan prior to approval for treatment. Dose volume histograms (DVH) and normal tissue constraint parameters specified below will be used to judge the plan quality and optimize PTV coverage with OAR sparing prior to approval.

Radiation will be delivered daily for 5 consecutive days with the exception of weekends and holidays. In instances where the radiation treatment week contains a holiday or scheduling availability is limited, two fractions of radiation may be given on the same day providing that the fractions are administered ≥ 6 hours apart (this is considered standard of care treatment).

Surgical resection of at least the primary tumor will follow within 12 weeks of completing radiation therapy. Surgical specimens will be sent to pathology for evaluation and for review by a multidisciplinary tumor board.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed sarcoma
* Primary or recurrent disease involving the abdomen or pelvis
* Resectable primary lesion
* Age ≥ 12 years old
* Karnofsky performance status (KPS) ≥ 70 or Eastern Cooperative Oncology Group (ECOG) 0-2
* If a woman is of childbearing potential, a negative serum or urine pregnancy test must be documented

Exclusion Criteria:

* Active treatment of a separate malignancy
* History of prior irradiation to the area targeted for treatment

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-05-30 (Actual); Primary Completion 2027-05-30 (Estimated); Study Completion 2028-05-26 (Estimated)

PRIMARY OUTCOMES:
Radiation morbidity at 2 years | At 2 years
  Evaluate the 2 year rate of grade ≥2 radiation morbidity, according to Common Terminology Criteria for Adverse Events (CTCAE), Version 5.0.

SECONDARY OUTCOMES:
Local Control | At 2 years
  Defined as freedom from radiographic progression of the treated site. It will be evaluated using CT and/or MRI of the abdomen and pelvis.
Regional Control | At 2 years
  Defined as freedom from radiographic progression in the abdomen or pelvis outside of the treated site. It will be evaluated using CT and/or MRI of the abdomen and pelvis.
Distant metastasis | At 2 years
Progression free survival | At 2 years
Overall survival | At 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- UCLA / Jonsson Comprehensive Cancer Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No